CLINICAL TRIAL: NCT02208531
Title: Transition to Scale of an Integrated Program of Nutritional Care and Psychosocial Stimulation to Improve Malnourished Children's Development in Bangladesh
Brief Title: Transition to Scale of Nutrition and Psychosocial Stimulation Program for Malnourished Children
Acronym: TTS Bangladesh
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: PR-13099
Record Dates: First submitted 2014-08-03; First posted 2014-08-05 (Estimated); Last update posted 2019-03-05 (Actual); Status verified 2018-08

CONDITIONS: Moderate and Severe Undernutrition
Keywords: Early Childhood Development (ECD); Psychosocial stimulation; Malnutrition; Bangladesh; Scaling up ECD
MeSH Terms: conditions — Lymphoma, Follicular; Malnutrition | interventions — Nutrition Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention)
- Psychosocial Stimulation and Nutritional Care (Experimental): Psychosocial Stimulation and Nutritional Care will be provided to malnourished children and their mothers every fortnight in the Community Clinics for one year.
  Interventions: Behavioral: Psychosocial Stimulation and Nutritional Care

INTERVENTIONS:
Behavioral: Psychosocial Stimulation and Nutritional Care — Psychosocial Stimulation and Nutritional Care will be provided to malnourished children and their mothers every fortnight in the Community Clinics for one year.
  Arms: Psychosocial Stimulation and Nutritional Care

SUMMARY:
We hypothesize that it is feasible to integrate a program of Nutritional Care and Pychosocial Stimulation into the Community Clinics in Bangladesh and thereby improve malnourished children's growth and development after a year of intervention.

DETAILED DESCRIPTION:
Over 200 million children <5 yrs do not reach their full potential due to poor nutrition and inadequate cognitive stimulation. Nutritional Care (NC) alone is insufficient to correct developmental deficit in malnourished children and psychosocial stimulation (PS) is also required.

Objectives:

1. Pilot two intervention methods and different delivery models of providing NC+PS to refine the intervention and identify any difficulties.
2. Conduct a cluster randomized controlled trial (CRCT) of NC+PS on malnourished children.
3. Pilot the feasibility of providing NC+PS to groups of mothers instead of individuals through a quasi-experimental design.

Methods: The study consists of 3 different sub-studies:

1. The pilot will be a qualitative study conducted in 10 Community Clinics (CCs) involving 40 children (aged 6-33 months) per CC. Mothers and children will attend the clinic every 2 weeks for an hour play session in groups of 2 or 6. We will explore different delivery models and assess problems through focus group discussions with parents and staff of the CCs.
2. For the CRCT we will survey all children aged 6-24 mo in 140 CCs to identify those malnourished. We will then randomize the CCs to NC+PS or control, randomly select 40 children from each CC and evaluate a random subsample of 6 children from each of the CCs using anthropometry, Bayley-III, Wolke's behavior rating and family care indicators (FCI) at baseline and endline.
3. The quasi experimental study will be conducted in 10 CCs randomized to group-intervention or control with 40 mothers and children per CC. Mothers will come to the CCs in groups of 6 with their children every fortnight. The children will be tested at the beginning and after 12 months using the same tools in the main study.

Outcome variable: The main outcomes are children's language, mental and psychomotor development measured on Bayley-III. In addition we expect improvements in FCI and mother's child rearing knowledge and practices. We will also conduct cost analysis and based on the success indicators, cost per successful outcome will be calculated from total cost of intervention program.

ELIGIBILITY:
Inclusion Criteria:

* Moderately and Severely malnourished children WAZ<-2SD
* Age: 6-24 months
* Both male and female children
* Living within 30 minutes walk from the Community Clinic
* Parents giving consent to participate in the study

Exclusion Criteria:

* Severe Acute Malnutrition with complications requiring close monitoring and/or hospitalization
* Severe clinical pallor
* Known chronic diseases like epilepsy, cerebral palsy, mental retardation
* Twin/multiple birth

Children with above exclusion criteria or those whose parents do not wish to sign the consent form will not be included in the evaluation sample but if they wish they will receive the stimulation.

Ages: 6 Months to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 6400 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2017-11-30 (Actual); Study Completion 2017-11-30 (Actual)

PRIMARY OUTCOMES:
Cognitive, Language and Motor Composite Scores | 12 months
  The outcomes are measured on Bayley-III test.
Anthropometry multiple measures, viz. Weight, length/height and head circumference | 12 months
  Children's weight, length/height and head circumference will be measured using standard methods.
Behaviour | 12 months
  The outcome is measured using Wolke's behaviour ratings during the Bayley-III test.

SECONDARY OUTCOMES:
Family Care Indicators | 12 months
  This outcome is measured by interviewing mothers of children about the quality of psychosocial stimulation at home.

CONTACTS AND LOCATIONS:
Locations (1):
- International Centre for Diarrhoeal Disease Research, Bangladesh, Dhaka, Bangladesh

REFERENCES:
- [Derived] Hossain SJ, Palmer T, Uddin Tipu SMM, Mehrin SF, Shiraji S, Hasan MI, Alam Bhuiyan MS, Salveen NE, Tofail F, Baker-Henningham H, Haghparast-Bidgoli H, Hamadani JD. Cost-effectiveness analysis of two integrated early childhood development programs into Bangladeshi primary health-care services. Lancet Reg Health Southeast Asia. 2025 Mar 28;35:100564. doi: 10.1016/j.lansea.2025.100564. eCollection 2025 Apr. PMID 40230446
- [Derived] Mehrin SF, Hasan MI, Tofail F, Shiraji S, Ridout D, Grantham-McGregor S, Hamadani JD, Baker-Henningham H. Integrating a Group-Based, Early Childhood Parenting Intervention Into Primary Health Care Services in Rural Bangladesh: A Cluster-Randomized Controlled Trial. Front Pediatr. 2022 Jun 10;10:886542. doi: 10.3389/fped.2022.886542. eCollection 2022. PMID 35783319
- [Derived] Hamadani JD, Mehrin SF, Tofail F, Hasan MI, Huda SN, Baker-Henningham H, Ridout D, Grantham-McGregor S. Integrating an early childhood development programme into Bangladeshi primary health-care services: an open-label, cluster-randomised controlled trial. Lancet Glob Health. 2019 Mar;7(3):e366-e375. doi: 10.1016/S2214-109X(18)30535-7. PMID 30784637